CLINICAL TRIAL: NCT07060079
Title: The Use of Entropy to Assess Sleep Disordered Breathing in Chronic Respiratory Disease
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 345082
Record Dates: First submitted 2025-06-26; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Bronchial Asthma; Bronchiectasis; ILD; COPD; OSAHS; OSA; Obesity Hypoventilation Syndrome (OHS)
Keywords: SDB; ILD; Entropy; bronchiectasis; COPD; asthma
MeSH Terms: conditions — Asthma; Bronchiectasis; Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Research is being conducted into chronic respiratory diseases, including chronic obstructive pulmonary disease (COPD), asthma, interstitial lung disease, and bronchiectasis. The investigation specifically focuses on sleep-disordered breathing (SDB) in individuals with chronic respiratory disease. SDB encompasses a range of conditions, the most common of which is obstructive sleep apnoea. In obstructive sleep apnoea, periodic pauses in breathing (apnoea) lead to reduced blood oxygen levels. To detect these events, patients typically undergo sleep studies that involve monitoring oxygen saturation, heart rate, and respiratory patterns during sleep. When chronic respiratory disease and SDB coexist, breathing disturbances during sleep may be exacerbated.

To identify SDB, sleep studies are commonly used to assess oxygen levels, heart rate, and breathing patterns. The objective of this research is to identify differences between patients with chronic respiratory diseases who have SDB and those who do not. This will be achieved by analysing sleep study data using a novel analytical approach. The aim is to determine whether this method can yield more detailed insights into the underlying pathophysiology of these conditions.

DETAILED DESCRIPTION:
Sleep is a complex and dynamic interplay between the brain and various physiological systems. Functions such as heart rate, respiration, and brain wave activity are regulated by intricate physiological mechanisms involving nonlinear interactions across multiple control centres operating on different time scales. It is increasingly recognized that a more accurate understanding of physiological outputs can be achieved through nonlinear analytical approaches, rather than traditional linear methods such as the standard deviation of the mean.

Among nonlinear techniques, entropy is one of the most widely used metrics for assessing the irregularity of physiological signals. For example, sample entropy is a method used to quantify regularity in time series data and has demonstrated the ability to distinguish between healthy and diseased individuals. In some cases, recordings from a simple finger pulse oximeter (measuring oxygen saturation (SpO₂)) may be sufficient to screen for sleep apnoea, potentially reducing the need for full cardiorespiratory polygraphy.

While nonlinear methods are well established in cardiovascular research, their application to respiratory signal analysis in obstructive sleep apnoea (OSA) remains limited. This analytical approach may offer deeper insights into complex physiological interactions-such as those between oxygen saturation and heart rate using relatively simple equipment.

The aim of this study is to investigate differences in entropy values between healthy individuals and patients with chronic respiratory diseases, both with and without coexisting sleep-disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥ 18years) with chronic respiratory disease with/without SDB.
* patients who have had previously negative studies as a control group.
* Subject is able to read, understand, and sign the informed consent form.
* Willing to sleep with portable monitoring devices.

Exclusion Criteria:

* Patients who are under 18 years of age at the time of the index study.
* Contraindications to the use of portable monitoring.
* Inability to give informed consent to take part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Royal Free Hospital in London over a period of 18 months. They will be approached during sleep or respiratory clinics attending and from an existing clinical database
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in respiratory signals entropy, oxygen saturation , and heart rate recorded using cardiorespiratory polygraphy during a 1-hour daytime and overnight sleep in healthy subjects and patients with chronic respiratory diseases with /without SDB. | 2 months
  High entropy value greater irregularity or complexity in the respiratory signal while low entropy value more regular, predictable, or uniform respiratory patterns.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El Shayeb M, Topfer LA, Stafinski T, Pawluk L, Menon D. Diagnostic accuracy of level 3 portable sleep tests versus level 1 polysomnography for sleep-disordered breathing: a systematic review and meta-analysis. CMAJ. 2014 Jan 7;186(1):E25-51. doi: 10.1503/cmaj.130952. Epub 2013 Nov 11. PMID 24218531
- [Result] Bhogal AS, Mani AR. Pattern Analysis of Oxygen Saturation Variability in Healthy Individuals: Entropy of Pulse Oximetry Signals Carries Information about Mean Oxygen Saturation. Front Physiol. 2017 Aug 2;8:555. doi: 10.3389/fphys.2017.00555. eCollection 2017. PMID 28824451